CLINICAL TRIAL: NCT01413347
Title: The Method to Reduce Displacement of Double-lumen Tube During Patient Positioning
Brief Title: The Method to Reduce Displacement of Double-lumen Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Hyon Bahk, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHBahk_DLT_pillow
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Double-lumen Tube Displacement

ARMS (2):
- pillow (Active Comparator): confirmation of double-lumen tube position with a head on a pillow
  Interventions: Procedure: pillow
- neutral (Experimental): confirmation of double-lumen tube position in neutral position of a head
  Interventions: Procedure: neutral

INTERVENTIONS:
Procedure: pillow — bronchoscopic confirmation of double-lumen tube position with a head on a pillow
  Arms: pillow
Procedure: neutral — bronchoscopic confirmation of double-lumen tube position in neutral position of a head
  Arms: neutral

SUMMARY:
The purpose of this study is to devise the method to reduce displacement of a left-sided double-lumen tube during patient positioning.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery that require the placement of left-sided double-lumen tubes

Exclusion Criteria:

* intraluminal lesion of left bronchus
* very distorted anatomy of tracheobronchial tree

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
tracheal displacement | up to 5 minutes

SECONDARY OUTCOMES:
bronchial displacement | up to 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Seo JH, Hong DM, Lee JM, Chung EJ, Bahk JH. Double-lumen tube placement with the patient in the supine position without a headrest minimizes displacement during lateral positioning. Can J Anaesth. 2012 May;59(5):437-41. doi: 10.1007/s12630-012-9679-7. Epub 2012 Feb 25. PMID 22368077